CLINICAL TRIAL: NCT05707455
Title: Hematological Factors and Iron Status in Aerobic Versus Anaerobic Training in Athletic Females: An Observational Study
Brief Title: Hematological Factors and Iron Status in Aerobic Versus Anaerobic Training in Athletic Females
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Assistant Professor, Cairo University
Other Study IDs: P.T.REC/012/004727
Record Dates: First submitted 2023-01-20; First posted 2023-02-01 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Sports Anemia
Keywords: Hematological factors; iron status; aerobic; anaerobic; athletic females; adolescence
MeSH Terms: interventions — Hematocrit; Erythrocyte Count; Erythrocyte Indices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aerobic group: long distance runners
  Interventions: Other: evaluating blood levels of hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin concentration, serum transferrin and serum ferritin.
- Anaerobic group: broad jumpers
  Interventions: Other: evaluating blood levels of hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin concentration, serum transferrin and serum ferritin.

INTERVENTIONS:
Other: evaluating blood levels of hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin concentration, serum transferrin and serum ferritin. — evaluating blood levels of hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin concentration, serum transferrin and serum ferritin.

SUMMARY:
This study aimed to evaluate the hematological factors and iron status in aerobic versus anaerobic training in athletic females.

DETAILED DESCRIPTION:
In both the short and long term, physical training causes iron status deterioration in sporty females. Nonetheless, little is known about the effect of different forms of exercise (aerobic versus anaerobic) on haematological variables and iron status in sporty females during adolescence. As a result, the purpose of this study was to compare the haematological variables and iron status in aerobic versus anaerobic exercise in adolescent female athletes. Another goal was to compare aerobic and anaerobic groups in terms of iron status classifications, such as normal iron status, iron deficiency with or without anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, virginal, nonsmoker, female athletes.
* Age from 16 to 19 years.
* Body mass index < 25 kg/m2.
* Having the same socio-economic level.
* Following a normal balanced nutrition.

Exclusion Criteria:

* Using any medical or hormonal therapy that might influence the iron status.
* Vegetarian athletes.
* Having menorrhagia or amenorrhea.
* Chronic inflammatory condition or existing infection.
* Diabetic, hypertensive or cardiac athletes.
* Haematological disease (with the exception of iron deficiency with or without anaemia).
* Having transfusion of blood.

Ages: 16 Years to 19 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: They were chosen via advertisement in local Cairo clubs.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Assessment of hemoglobin (Hb) | 2 months
  Blood samples were collected between 8:00 and 9:00 a.m. after an overnight fast and time of relaxation. The athletic girls were asked to refrain from exercising the day before sample. Blood was taken from the antecubital vein and placed in one EDTA tube and one beads tube for serum separation. An automatic cell counter (Sysmex XS 1000, Japan) was used to measure hemoglobin (Hb).
Assessment of hematocrit (Hct) | 2 months
  Blood samples were collected between 8:00 and 9:00 a.m. after an overnight fast and time of relaxation. The athletic girls were asked to refrain from exercising the day before sample. Blood was taken from the antecubital vein and placed in one EDTA tube and one beads tube for serum separation. An automatic cell counter (Sysmex XS 1000, Japan) was used to measure hematocrit (Hct).
Assessment of red blood cell (RBC) count | 2 months
  Blood samples were collected between 8:00 and 9:00 a.m. after an overnight fast and time of relaxation. The athletic girls were asked to refrain from exercising the day before sample. Blood was taken from the antecubital vein and placed in one EDTA tube and one beads tube for serum separation. An automatic cell counter (Sysmex XS 1000, Japan) was used to measure red blood cell (RBC) count.
Assessment of mean corpuscular volume (MCV) | 2 months
  Blood samples were collected between 8:00 and 9:00 a.m. after an overnight fast and time of relaxation. The athletic girls were asked to refrain from exercising the day before sample. Blood was taken from the antecubital vein and placed in one EDTA tube and one beads tube for serum separation. An automatic cell counter (Sysmex XS 1000, Japan) was used to measure mean corpuscular volume (MCV).
Assessment of mean corpuscular hemoglobin concentration (MCHC) | 2 months
  Blood samples were collected between 8:00 and 9:00 a.m. after an overnight fast and time of relaxation. The athletic girls were asked to refrain from exercising the day before sample. Blood was taken from the antecubital vein and placed in one EDTA tube and one beads tube for serum separation. An automatic cell counter (Sysmex XS 1000, Japan) was used to measure mean corpuscular hemoglobin concentration (MCHC).
Assessment of serum transferrin | 2 months
  Blood samples were collected between 8:00 and 9:00 a.m. after an overnight fast and time of relaxation. The athletic girls were asked to refrain from exercising the day before sample. Blood was taken from the antecubital vein and placed in one EDTA tube and one beads tube for serum separation. The serum sample was centrifuged, and the serum transferrin was measured using COBAS Integra 400 plus, Switzerland.
Assessment of serum ferritin | 2 months
  Blood samples were collected between 8:00 and 9:00 a.m. after an overnight fast and time of relaxation. The athletic girls were asked to refrain from exercising the day before sample. Blood was taken from the antecubital vein and placed in one EDTA tube and one beads tube for serum separation. The serum sample was centrifuged, and the serum ferritin was measured using ADVIA Centaur XPT, Germany.

SECONDARY OUTCOMES:
Anthropometric measures | 2 months
  A weight-height scale was used to assess the weight (Kg) and height (m) for each female athlete in the two groups. The body mass index (BMI) was then calculated by dividing the weight by the height squared (Kg/m2).
Assessment of participation age to sport | 2 months
  Each female athlete was asked about her age of participation to sport to assess her training profile.
Assessment of number of hours of training per week | 2 months
  Each female athlete was asked about the number of hours of training per week to assess her training profile.
Assessment of training experience | 2 months
  The training experience in years was calculated by subtracting the female athlete's age of participation to training from her chronological age.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Osman, Assis. Prof., Principal Investigator — Physical Therapy for Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Local clubs, Cairo, Egypt